CLINICAL TRIAL: NCT07208071
Title: Application of Augmented Reality for Point of Care Ultrasound-Guided Procedures
Brief Title: Investigating the Utility of Augmented Reality Assistance for Ultrasound-Guided Vascular Access
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jeffrey Coote, Pediatric Critical Care Fellow, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300014090; UAB (Other: UAB)
Record Dates: First submitted 2025-09-19; First posted 2025-10-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Vascular Access
Keywords: Augmented reality; ultrasound-guided vascular access

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Providers will not use augmented reality assistance when performing ultrasound-guided vascular access for this arm of the study
- AR Arm (Experimental): Providers will use augmented reality assistance when obtaining ultrasound-guided vascular access
  Interventions: Other: Augmented reality headset use

INTERVENTIONS:
Other: Augmented reality headset use — Use of a Microsoft HoloLens 2 headset with augmented reality assistance
  Arms: AR Arm

SUMMARY:
This study will investigate the benefits of augmented reality assistance on ultrasound-guided vascular access. Using the Microsoft HoloLens 2 headset, the investigators will study the benefits of augmented reality technology as a tool for improving the success rate, efficiency, and ease of access for peripheral venous catheters, peripherally inserted central venous catheters, and central venous catheters.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring ultrasound-guided vascular access

Exclusion Criteria:

* Age less than 5 years old
* Need for urgent vascular access

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Successful vascular access as indicated by blood return from the blood vessel and advancement of guide wire | Up to 30 minutes

SECONDARY OUTCOMES:
Number of needle sticks required for successful vascular access | Up to 30 minutes
Time required for successful vascular access | Up to 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Saruwatari MS, Nguyen TN, Talari HF, Matisoff AJ, Sharma KV, Donoho KG, Basu S, Dwivedi P, Bost JE, Shekhar R. Assessing the Effect of Augmented Reality on Procedural Outcomes During Ultrasound-Guided Vascular Access. Ultrasound Med Biol. 2023 Nov;49(11):2346-2353. doi: 10.1016/j.ultrasmedbio.2023.07.011. Epub 2023 Aug 11. PMID 37573178